CLINICAL TRIAL: NCT03962088
Title: Timing To Minimally Invasive Surgery After Neoadjuvant Chemoradiotherapy For Rectal Cancer: A Multicenter Randomized Controlled Trial - Biomarkers SubStudy
Brief Title: Timisnar - Biomarkers Substudy (Timisnar-mirna)
Acronym: TiMiSNAR-miRNA
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Principal Investigator, Igor Monsellato, Principal Investigator, Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria
Other Study IDs: A19
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Total RNA, including miRNAs, are isolated using a commercial kit (miRNeasy Mini Kit, Qiagen, Hilden, Germany) according to the manufacturer's instructions. The RNA concentration is assessed using a spectrophotometer. The RNA results adequate for mRNA expression whenever its concentration is ≥30 ng/μL and its quality is acceptable if the ratio between the value of the absorbance (A) at 260 nm and the absorbance at 280 nm is ≥1.8, and the ratio between the value of absorbance (A) at 260 nm and the one at 230 nm is ≥2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: miRNA — 15 ml of whole blood samples are collected in Vacutainer tubes with spray-coated K2EDTA and stored at room temperature. To minimize the hemolysis and nucleic acids degradation, plasma separation undergoes within 2 h.
  Within 1 h, tubes are subjected to a first centrifugation step at 2200 x g and room temperature for 15 min. Plasma supernatants are transferred to 15 mL tubes, carefully avoiding contact with the lymphocytic ring, and tubes are centrifuged a second time at 3000 x g and RT for 10 min to remove cellular debris.
  Plasma samples are then collected into 1.5 mL cryovials and all the aliquots are stored at -80 °C.

SUMMARY:
Neoadjuvant chemoradiotherapy (nCHT) followed by surgery is the mainstay treatment for locally advanced rectal cancer, leading to significant decrease in tumor size (downsizing) and a shift towards earlier disease stage in the primary tumor and lymph nodes (downstaging). Extensive histopathological work-up of the tumor specimen after surgery including tumor regression grading (TRG) and lymph node status (ypN) helped to visualize individual tumor sensitivity to CRT retrospectively. Since the response to nCHT is heterogeneous, however, valid biomarkers are needed to monitor tumor response. A relevant number of studies aimed to identify molecular markers retrieved from tumor tissue while the relevance of blood-based biomarkers is less stringent assessed.

As a potential alternative to CEA and ctDNA, microRNAs (miRNAs) are currently under investigation to serve as blood-based biomarkers. miRNAs are small, noncoding RNAs that regulate gene expression by post-transcriptional mRNA binding, which promotes the destabilization of target miRNAs. The target specificity of miRNAs is largely predetermined by their so-called "seed-sequence" (containing nucleotides at position 2-7 of the miRNA). They are highly conserved between species, stable and easy detectable even in small concentrations. They have been widely analyzed in physiological and pathological processes, and their expression is tissue specific.

DETAILED DESCRIPTION:
Neoadjuvant chemoradiotherapy (nCHT) followed by surgery is the mainstay treatment for locally advanced rectal cancer, leading to significant decrease in tumor size (downsizing) and a shift towards earlier disease stage in the primary tumor and lymph nodes (downstaging). Extensive histopathological work-up of the tumor specimen after surgery including tumor regression grading (TRG) and lymph node status (ypN) helped to visualize individual tumor sensitivity to CRT retrospectively. Since the response to nCHT is heterogeneous, however, valid biomarkers are needed to monitor tumor response. A relevant number of studies aimed to identify molecular markers retrieved from tumor tissue while the relevance of blood-based biomarkers is less stringent assessed.

Blood samples, i.e. Liquid Biopsy, however, offer several advantages:

1. Taking blood samples is less invasive, less expensive, easy to schedule, and nearly without any severe complications.
2. Blood samples are a source of fresh DNA and RNA, without modifications due to preservatives; especially in the case of rectal cancer, beyond intratumoral heterogeneity, tumor biopsies are in general accompanied by normal, adenomatous or stromal tissue. This contamination may affect results of molecular analyses
3. Investigating blood from patients can account for molecular heterogeneity and surrogate for tumor burden since tumor-derived fragments or biomarkers are collected from all tumor cells in a patients' body through circulation.
4. Liquid biopsy may offer both the possibility of dynamic monitoring under treatment and the possibility to assess disease activity even after pathologic complete response (pCR) or after resection of the tumor when no tissue is left for molecular analyses.

In clinical routines, to date, carcinoembryonic antigen (CEA) is established as a colorectal cancer (CRC) related tumor marker but is not recommended as a screening test for colorectal cancer. First, normal levels of CEA do not exclude the possibility of a colorectal cancer. Second, an elevated CEA is not categorically associated with CRC, or in the period of follow-up with disease progression. Circulating tumor DNA (ctDNA) represents nowadays, the main approach to monitor tumor burden and therapy resistance, to evaluate the presence of residual disease after potentially curative treatment and to monitor disease recurrence with high sensitivity and specificity.

As a potential alternative to CEA and ctDNA, microRNAs (miRNAs) are currently under investigation to serve as blood-based biomarkers. miRNAs are small, noncoding RNAs that regulate gene expression by post-transcriptional mRNA binding, which promotes the destabilization of target miRNAs. The target specificity of miRNAs is largely predetermined by their so-called "seed-sequence" (containing nucleotides at position 2-7 of the miRNA). They are highly conserved between species, stable and easy detectable even in small concentrations. They have been widely analyzed in physiological and pathological processes, and their expression is tissue specific.

To date, no screening approach to identify relevant miRNAs as biomarkers in blood of patients with rectal cancer was undertaken.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* cT3/4N0/+M0 confirmed on CT-scan, MRI (stratification for T3a-b-c-d)
* Histologically-proven adenocarcinoma of the rectum
* Eligible for a resective surgery with TME
* Eligible for chemoradiation treatment

Exclusion Criteria:

* Metastatic disease
* Squamous carcinoma of the anal canal
* Unable to complete neoadjuvant treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All included patients in the TiMiSNAR Trial (already approved by local Ethical Committees on 8/5/2018 - NCT3465982) are supposed to undergo blood collection at the time of diagnosis, after neoadjuvant treatment, after 1 month from surgery and after adjuvant chemotherapy whenever indicated.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in expression levels of plasma miRNA | 5 years
  the association of variation between preneoadjuvant and postneoadjuvant expression levels of miRNA with pCR

SECONDARY OUTCOMES:
miRNA expression and surgery | 5 years
  changes in expression levels of miRNA following complete surgical resection with disease-free survival
miRNA expression and surveillance | 5 years
  the relation between changes in miRNA during surveillance and tumor relapse

CONTACTS AND LOCATIONS:
Locations (1):
- SS. Antonio e Biagio e Cesare Arrigo, Alessandria, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yu J, Li N, Wang X, Ren H, Wang W, Wang S, Song Y, Liu Y, Li Y, Zhou X, Luo A, Liu Z, Jin J. Circulating serum microRNA-345 correlates with unfavorable pathological response to preoperative chemoradiotherapy in locally advanced rectal cancer. Oncotarget. 2016 Sep 27;7(39):64233-64243. doi: 10.18632/oncotarget.11649. PMID 27572313
- [Result] Dayde D, Tanaka I, Jain R, Tai MC, Taguchi A. Predictive and Prognostic Molecular Biomarkers for Response to Neoadjuvant Chemoradiation in Rectal Cancer. Int J Mol Sci. 2017 Mar 7;18(3):573. doi: 10.3390/ijms18030573. PMID 28272347
- [Result] Rampazzo E, Del Bianco P, Bertorelle R, Boso C, Perin A, Spiro G, Bergamo F, Belluco C, Buonadonna A, Palazzari E, Lonardi S, De Paoli A, Pucciarelli S, De Rossi A. The predictive and prognostic potential of plasma telomerase reverse transcriptase (TERT) RNA in rectal cancer patients. Br J Cancer. 2018 Mar 20;118(6):878-886. doi: 10.1038/bjc.2017.492. Epub 2018 Feb 15. PMID 29449673
- [Result] Augestad KM, Merok MA, Ignatovic D. Tailored Treatment of Colorectal Cancer: Surgical, Molecular, and Genetic Considerations. Clin Med Insights Oncol. 2017 Feb 16;11:1179554917690766. doi: 10.1177/1179554917690766. eCollection 2017. PMID 28469509
- [Result] Drebber U, Lay M, Wedemeyer I, Vallbohmer D, Bollschweiler E, Brabender J, Monig SP, Holscher AH, Dienes HP, Odenthal M. Altered levels of the onco-microRNA 21 and the tumor-supressor microRNAs 143 and 145 in advanced rectal cancer indicate successful neoadjuvant chemoradiotherapy. Int J Oncol. 2011 Aug;39(2):409-15. doi: 10.3892/ijo.2011.1036. Epub 2011 May 10. PMID 21567082
- [Result] Della Vittoria Scarpati G, Falcetta F, Carlomagno C, Ubezio P, Marchini S, De Stefano A, Singh VK, D'Incalci M, De Placido S, Pepe S. A specific miRNA signature correlates with complete pathological response to neoadjuvant chemoradiotherapy in locally advanced rectal cancer. Int J Radiat Oncol Biol Phys. 2012 Jul 15;83(4):1113-9. doi: 10.1016/j.ijrobp.2011.09.030. Epub 2011 Dec 13. PMID 22172905
- [Derived] Monsellato I, Garibaldi E, Cassinotti E, Baldari L, Boni L, Elmore U, Delpini R, Rosati R, Perinotti R, Alongi F, Bertocchi E, Gori S, Ruffo G, Pernazza G, Pulighe F, De Nisco C, Morpurgo E, Contardo T, Mammano E, Perna F, Menegatti B, Coratti A, Buccianti P, Balestri R, Ceccarelli C, Cavaliere D, Solaini L, Ercolani G, Traverso E, Fusco V, Torri V, Orecchia S. Expression levels of circulating miRNAs as biomarkers during multimodal treatment of rectal cancer - TiMiSNAR-mirna: a substudy of the TiMiSNAR Trial (NCT03962088). Trials. 2020 Jul 25;21(1):678. doi: 10.1186/s13063-020-04568-9. PMID 32711544
- See also: Official site of the study — https://mirna.timisnar.it